CLINICAL TRIAL: NCT01813240
Title: Prevention of Imminent Paralysis Following Spinal Cord Trauma or Ischemia by Minocycline: A Multi-center Study in Israel With IDF Primary Care Involvement
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Benjamin Drenger, Associate Professor of Anesthesia, Director, Orthopedic Anesthesia,, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0727-11-HMO
Record Dates: First submitted 2013-03-11; First posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Spinal Tumors, Trauma Patients, Minocycline.
MeSH Terms: conditions — Spinal Cord Neoplasms; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Minocycline, Spinal Tumor patients, quality of life (Experimental)
  Interventions: Drug: Minocycline
- Minocycline, Trauma patuents, quality of life (Experimental)
  Interventions: Drug: Minocycline
- Placebo, Trauma patients, quality of life (Placebo Comparator)
  Interventions: Drug: placebo
- Placebo, Spinal cord tumors, quality of life (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Minocycline
  Arms: Minocycline, Spinal Tumor patients, quality of life; Minocycline, Trauma patuents, quality of life
Drug: placebo
  Arms: Placebo, Spinal cord tumors, quality of life; Placebo, Trauma patients, quality of life

SUMMARY:
Spinal cord trauma and the consequent paraplegia are possibly among the most devastating injuries in soldiers and during spine surgery, and are significant in the medical, social and financial aspects. Limited mobility, the need for assistance in all human activities, shame, and many medical complications related directly to the neural deficits make paraplegia an important target for prevention. Our study will evaluate the efficacy of Minocycline in two different groups:

1. Minimizing the neurological damage among trauma patients.
2. Preventing neurological damage through operation in spinal tumors patients.

2.OBJECTIVES

The primary objectives of the trial are to determine:

1. Efficacy of administrating minocycline in minimizing the neurological damage among acute spinal cord injury patients and spinal cord tumors (primary and metastases) patients?
2. Efficacy of administrating minocycline at changing the natural history and rehabilitation of spinal cord trauma patients.
3. Safety of applying minocycline in spinal cord injuries patients and spinal cord tumors?

ELIGIBILITY:
Inclusion Criteria:

Trauma patients with incomplete spinal cord syndromes related to fractures, dislocations, blunt trauma (central cord syndrome).

1. Inclusion Criteria:
2. Patients with incomplete spinal cord syndromes related to fractures, dislocations, blunt trauma (central cord syndrome).
3. Ages: 18 to 65
4. Males - including those involved in active military duty.
5. Females - of child-bearing potential who have a negative pregnancy test (hCG urine) within 72 hours of informed consent. Pregnant women will be excluded from the study.

Exclusion Criteria:

1. Complete cord transection, severe head injury, coma, or other disease of the CNS, and spinal injury diagnosed later than 24 hours.
2. Pregnant women (minocycline can cause fetal harm) and children.
3. Lower extremity fractures, mildly reduced consciousness and frail cognitive status will not be considered for exclusion.
4. Patients who will not be enrolled will be listed and reason for non inclusion will be recorded.

Spinal tumors:

Inclusion Criteria:

1. Intrathecal extramedullary tumors, vertebral metastases or primary vertebral tumors causing cord compression with or without incomplete cord syndrome.

Exclusion criteria:

1.Intramedullary tumors or tumors causing complete cord syndrome

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of administrating minocycline in minimizing the neurological damage among acute spinal cord injury patients and spinal cord tumors (primary and metastases) patients | six months
  The Efficacy will be evaluated using the following measures:
  1. ASIA SCORE - We will compare the results before administrating the study medication and after six months of follow up. The ASIA score will be the Primary Efficacy Endpoint.
  2. The Spinal Cord Independence Measure and Functional Independence Measure outcome scales.
  3. Objective reduction in lesion size by imaging modalities

SECONDARY OUTCOMES:
Efficacy of administrating minocycline at changing the natural history and rehabilitation of spinal cord trauma patients. | six months
  The Efficacy will be evaluated using the following measures:
  1. ASIA SCORE - We will compare the results before administrating the study medication and after six months of follow up. The ASIA score will be the Primary Efficacy Endpoint.
  2. The Spinal Cord Independence Measure and Functional Independence Measure outcome scales.
  3. Objective reduction in lesion size by imaging modalities
Safety of applying minocycline in spinal cord injuries patients and spinal cord tumors? | six months
  Safety will be evaluated in a descriptive manner by recording all adverse events in the patient population by number and severity.
  The study will evaluate safety by assessing:
  * Procedure related adverse events:
  * General adverse events: Adverse events not only directly related to the procedure, such as: complications related to anesthesia, hospitalization, or other general adverse events of unknown cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel